CLINICAL TRIAL: NCT06016075
Title: Investigation of Differential Biology of Benign and Malignant Renal Masses Using Advanced Magnetic Resonance Imaging Techniques
Acronym: IBM-Renal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Ines Horvat-Menih, Doctor, University of Cambridge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Radiology, Uni of Cambridge; 22/EE/0136 (Registry Identifier: Health Research Authority, East of England - Cambridge East Research Ethics Committee); 314155 (Registry Identifier: Integrated Research Application System)
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyperpolarised MRI (Other): Hyperpolarised 13C-pyruvate injection while laying in the MRI scanner. Non-radioactive, no risk, approved for use in humans.
  Interventions: Device: Hyperpolarised MRI
- Sodium MRI (Other): MRI procedure as a regular MRI scan, the only change is us using a different sort of equipment so we are able to detect sodium.
  Interventions: Device: Sodium MRI
- Deuterium metabolic imaging (DMI) MRI (Other): Drink of a sugar drink 90min before the MRI scan. Non-radioactive, no risk, approved for use in humans.
  Interventions: Device: Deuterium metabolic imaging (DMI) MRI

INTERVENTIONS:
Device: Hyperpolarised MRI — Hyperpolarised 13C-pyruvate injection while laying in the MRI scanner. Non-radioactive, no risk, approved for use in humans.
  Arms: Hyperpolarised MRI
Device: Sodium MRI — MRI procedure as a regular MRI scan, the only change is us using a different sort of equipment so we are able to detect sodium.
  Arms: Sodium MRI
Device: Deuterium metabolic imaging (DMI) MRI — Drink of a sugar drink 90min before the MRI scan. Non-radioactive, no risk, approved for use in humans.
  Arms: Deuterium metabolic imaging (DMI) MRI

SUMMARY:
The aim of this study is to develop techniques for non-invasive imaging of biology in participants with benign or malignant renal masses based on the novel scanning MRI techniques, including recently invented Hyperpolarised MRI, deuterium metabolic imaging and sodium MRI. This imaging study will: 1) acquire imaging data from human tissues following the injection of hyperpolarised 13C pyruvate and use 13C-MRI to monitor changes in the ratio of 13C-lactate to 13C-pyruvate; 2) acquire imaging data from human tissues using Sodium MRI or 3) acquire imaging data from human tissues following the oral consumable of deuterated glucose. Data acquired during this physiological study will be used to optimise future imaging protocols.In the UK and possibly in other countries, there are some patients with renal masses that are over treated or undergo unnecessary procedures such as surgery or biopsies, as they are thought to have a malignant tumour or a more aggressive tumour but after the procedure it is found that the mass was benign. The aim of this study is to determine whether one or all of these imaging techniques can differentiate between benign and malignant renal masses with the view to developing the techniques further and hopefully reducing the need for over treatment or unnecessary procedures in patients with benign masses.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Able to and provide written informed consent to participate
* If female, postmenopausal or if women of child bearing potential (WOCBP) using a suitable contraception
* If male, using a suitable contraceptive method for the duration of the study
* Radiologically suspected or pathologically confirmed benign or malignant renal masses, as determined by standard clinical practice
* Capable of undergoing a minimum of one study visit

Exclusion Criteria:

* Contraindication or inability to tolerate MRI
* Pregnant or actively breast-feeding woman
* If using an intrauterine contraceptive device (IUCD) as a method of contraception the device should be MRI safe at 3 T (researcher to confirm)
* Clinically significant cardiac, pulmonary or neurological diseases as determined by the investigators
* Laboratory abnormalities that may impact on the study results
* Any other significant medical or psychiatric history rendering the subject ineligible as deemed by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
LAC/PYR ratio | 1 year
  LAC/PYR ratio in renal tumours, which is a quantitative measure of conversion from pyruvate to lactate in the tissue of interest.
Total Sodium Concentration | 1 year
  Total Sodium Concentration - in renal tumours
Technical development of DMI in the abdomen | 1 year
  Detection of metabolites within the DMI spectrum in the abdomen is limited by large lipid peaks and variability of tissues. Therefore, this work will aim to improve acquisition and processing methods to develop abdominal DMI with the hope to evaluate lactate across renal tumour subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdia A Gallagher, MD PhD, Principal Investigator — Principal Investigator
Locations (1):
- University Department of Radiology, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horvat-Menih I, McLean MA, Zamora-Morales MJ, Wylot M, Kaggie J, Khan AS, Gill AB, Duarte J, Locke MJ, Mendichovszky I, Li H, Priest AN, Warren AY, Welsh SJ, Jones JO, Armitage JN, Mitchell TJ, Stewart GD, Gallagher FA. Multiarm, non-randomised, single-centre feasibility study-investigation of the differential biology between benign and malignant renal masses using advanced magnetic resonance imaging techniques (IBM-Renal): protocol. BMJ Open. 2024 Oct 26;14(10):e083980. doi: 10.1136/bmjopen-2024-083980. PMID 39461869